CLINICAL TRIAL: NCT03654443
Title: Greek Validation of the Critical-Care Pain Observation Tool (CPOT) in the Intensive Care Unit Setting
Brief Title: Validation of the Critical-Care Pain Observation Tool (CPOT) in the Greek Population
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is currently suspended due to the COVID19 crisis
Sponsor: Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Georgia Micha, Principal Investigator, Anaesthesiologist, MD, MSc, PhD, Saint Savvas Anticancer Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: StSavvasAH
Record Dates: First submitted 2018-06-16; First posted 2018-08-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pain; Intensive Care Units
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the two observers are aware of the study group and none of the rest of the study team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Painful stimulus (Experimental): The CPOT tool is administered in a crossover manner in Group one prior to a painful stimulus (IT0), during the painful stimulus (IT1) and soon afterwards (IT2)
  Interventions: Diagnostic Test: Critical care pain observation tool
- Group Non-painful stimulus (Experimental): The CPOT tool is administered in a crossover manner in Group one prior to a non-painful stimulus (IIT0), during the painful stimulus (IIT1) and soon afterwards (IIT2)
  Interventions: Diagnostic Test: Critical care pain observation tool

INTERVENTIONS:
Diagnostic Test: Critical care pain observation tool — The CPOT tool is administered in a crossover manner by two study observers

SUMMARY:
The aim of this study is to validate the Critical-Care Pain Observation Tool (CPOT) in the setting of the Intensive care unit (ICU). Prior to patient recruitment the tool will be translated by the method of translation-back translation by Greek and English native speakers. The tool will be administered to patients who are admitted into the ICU.

DETAILED DESCRIPTION:
The aim of this study is to validate the Critical-Care Pain Observation Tool (CPOT) in the setting of the Intensive care unit (ICU). Prior to patient recruitment the tool will be translated by the method of translation-back translation by Greek and English native speakers. The study is designed as a prospective randomized crossover clinical trial. Patients will be randomly allocated into two study groups. In Group I the CPOT tool is administered prior to a painful stimulus (ITime0), during the painful stimulus (ITime1) and soon afterwards (ITime2).In Group II the CPOT tool is administered prior to a non painful stimulus(IITime0), during a non-painful stimulus (IITime1) and soon afterwards (IITime2). After these trials the patients in the two groups will crossover into the other group and the whole process will be repeated. The painful stimulus is set to be the passive turning of the patient into the bed and the non painful stimulus is the cleaning of the arm or leg. 20 minutes afterwards the CPOT tool is administered once again in both groups in order to obtain the values when there is no stimulus (ITime3). The tool is administered by two trained members of the study team in a blind manner. Both of the observers administer the tool at the same time but one of them is positioned in the ward of the patient and the other one behind a curtain with no contact with the observer but only with the patient and the monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the ICU
* Age> 18 years old
* No hearing or visual deficit
* No contraindication to body repositioning

Exclusion Criteria:

* Patients with neurological deficit
* Patients administered with neuromuscular blocking agents
* Patients with motor or sensory deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool (Critical Care Pain Observation Tool) is administered 1 minute prior to a painful stimulus (ITime0) which is set to be the patient's bed repositioning
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool(Critical Care Pain Observation Tool) is administered 10 seconds after a painful stimulus (ITime1) which is set to be the patient's bed repositioning
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool(Critical Care Pain Observation Tool) is administered 1 minute after a painful stimulus (ITime2) which is set to be the patient's bed repositioning
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool (Critical Care Pain Observation Tool)is administered 20 minutes after a painful stimulus (ITime3) which is set to be the patient's bed repositioning
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool (Critical Care Pain Observation Tool)is administered 1 minute prior to a non painful stimulus (IITime0) which is set to be the patient's blood pressure measurement
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool(Critical Care Pain Observation Tool) is administered 10 seconds after a non painful stimulus (IITime1) which is set to be the patient's blood pressure measurement
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.
Greek validation of the CPOT tool (Critical Care Pain Observation Tool) in the ICU patients | The CPOT tool (Critical Care Pain Observation Tool)is administered 1 minute after a painful stimulus (IITime2) which is set to be the patient's blood pressure measurement
  Validation of the Greek version of the CPOT tool (Critical Care Pain Observation Tool) for assessing the pain in the intensive care unit patients.Maximum score 8 points.For those patients with a CPOT score of ≤ 2:There is likely minimal to no pain present.For those patients with a CPOT score of >2:There is a medium to severe level of pain.

SECONDARY OUTCOMES:
Correlation of physiological parameters to CPOT tool (Critical Care Pain Observation Tool) values | The recordings will be performed 1 minute before, 10 seconds after, 1 minute after and 20 minutes after a painful and a non painful stimulus
  Physiological parameters as mean arterial blood pressure (MAP in mmHg) will be recorded in all patients. In order to calculate the mean arterial pressure, systolic and diastolic pressures will be recorded in the time periods of the assessment.
Correlation of numeric pain rating scale (NPRS) to CPOT tool (Critical Care Pain Observation Tool)values | The recordings will be performed 1 minute before, 10 seconds after, 1 minute after and 20 minutes after a painful and a non painful stimulus
  NPRS scale (0 equals no pain and 10 equals maximum pain possible)will be performed in all patients that are able to communicate in order to correlate the results with those of the CPOT tool
Correlation of physiological parameters to CPOT tool(Critical Care Pain Observation Tool) values | The recordings will be performed 1 minute before, 10 seconds after, 1 minute after and 20 minutes after a painful and a non painful stimulus
  Physiological parameters as heart rate will be recorded in all patients.
Correlation of physiological parameters to CPOT tool (Critical Care Pain Observation Tool)values | The recordings will be performed 1 minute before, 10 seconds after, 1 minute after and 20 minutes after a painful and a non painful stimulus
  Physiological parameters as respiratory rate will be recorded in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Micha, MD, MSc, PhD, Principal Investigator — Saint Savvas Anticancer Hospital of Athens
Locations (1):
- Saint Savvas Anticancer Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gelinas C, Fillion L, Puntillo KA. Item selection and content validity of the Critical-Care Pain Observation Tool for non-verbal adults. J Adv Nurs. 2009 Jan;65(1):203-16. doi: 10.1111/j.1365-2648.2008.04847.x. Epub 2008 Nov 15. PMID 19032510
- [Background] Kanji S, MacPhee H, Singh A, Johanson C, Fairbairn J, Lloyd T, MacLean R, Rosenberg E. Validation of the Critical Care Pain Observation Tool in Critically Ill Patients With Delirium: A Prospective Cohort Study. Crit Care Med. 2016 May;44(5):943-7. doi: 10.1097/CCM.0000000000001522. PMID 26783859